CLINICAL TRIAL: NCT03084627
Title: Evaluation of the Efficiency of Tailored Dietary Advice in Improving the Nutrient Adequacy of the Diet of French Pregnant Women
Acronym: MONCAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: AgroParisTech, INRA, Université Paris-Saclay (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MONCAP
Record Dates: First submitted 2017-03-01; First posted 2017-03-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy
Keywords: tailored dietary advice; nutrient adequacy; dietary modifications

STUDY DESIGN:
Who Masked: Participant
Masking Description: volunteers (single masking)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generic dietary advice for pregnancy (No Intervention)
- Generic dietary advice for pregnancy + Tailored dietary advice (Experimental)
  Interventions: Behavioral: Tailored dietary advice

INTERVENTIONS:
Behavioral: Tailored dietary advice — The nutrient adequacy of the diet of each patient will be evaluated, at baseline, by a diet quality index: the PANDiet. Then, tailored dietary advice aiming at improving the nutrient adequacy of the diet will be generated for each patient in the arm #2. Patients will choose 3 tailored dietary advices among 3 options during three appointments with a research project team member (the first in person and the second and the third by phone). Each appointment will be spaced of 2 weeks. In total, each patient in the arm #2 will choose nine tailored dietary advice. Tailored dietary advices are of two kinds: substitution of a consumed food item by a food item in the same food subgroup or modification of the consumed amount (increase or decrease) of a food item. Tailored dietary advices cannot generate an increase of more than 190 kcal or a decrease as compared to the observed energy intake.
  Arms: Generic dietary advice for pregnancy + Tailored dietary advice

SUMMARY:
Pregnancy is associated with an increase in nutrient requirements. During this period, women would be keener on adopting healthier behaviors. Thus, pregnancy represents an opportunity to improve the nutrient adequacy of the diet of mothers-to-be. This study is a randomized controlled trial, which aims at evaluating the efficiency of a tailored dietary advice tool in improving the nutrient adequacy of the diet of pregnant women, as measured by the PANDiet. Eighty pregnant women will be included in the study and randomized either in the "control" group, or in the "intervention" group. The control group will receive generic dietary advice based on a booklet edited by the French Institute for Health Promotion and Health Education (INPES). The intervention group will receive the same generic dietary advice plus tailored dietary advice to improve the nutrient adequacy of their observed diets. Dietary intakes will be evaluated online using a 3 days food record, at baseline and 6 weeks after patients received the booklet and/or the first tailored dietary advice. Thus, the nutrient adequacy of the diet could be evaluated before and after the intervention in both groups.

The dietary follow-up for one patient will last 12 weeks only, but data will be collected at delivery.

"Moreover, after, the 12-week dietary follow-up and before their deliveries, 10 participants (5 by group) will be contacted to participate in a qualitative interview. This interview will aim at understanding barriers and motivators to implement dietary advice (generic and/or tailored) in the diet of pregnant women in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Pregnant (between 10 and 24 amenorrhea weeks)
* Aged from 18 to 40
* BMI between 18.5 and 25 kg/m²
* Singleton pregnancy
* Fluently speaking, writing and reading of French
* Having a daily internet access, a personal email address and phone number
* Benefiting from the French Health Coverage
* Not suffering from a gestational diabetes during this pregnancy or a previous pregnancy
* Not being on a specific diet for medical purpose
* Not suffering from major food allergies

Exclusion Criteria:

* Diagnosis of a gestational diabetes during the 12 weeks of the study
* Diagnosis of a pathology that would require diet modifications during the 12 weeks of the study.
* Abortion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female because it's a study about pregnancy
Enrollment: 80 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The improvement in the PANDiet, a diet quality index which has been adapted to pregnancy. | Week 2 Week 3 week 11 week 12

SECONDARY OUTCOMES:
frequency of dietary advice applied | week 12
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean François HUNEAU, Professor, Study Director — UMR Physiologie de la Nutrition et du Comportement Alimentaire INRA/AgroParisTech; Elie AZRIA, MD, Principal Investigator — Groupe Hospitalier Paris St Joseph; Clelia BIANCHI, PhD student, Study Director — UMR Physiologie de la Nutrition et du Comportement Alimentaire INRA/AgroParisTech
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No